CLINICAL TRIAL: NCT02782494
Title: Comparing Consistency of QuantiFERON-TB Gold Plus and QuantiFERON-TB Gold for Latent Tuberculosis in Dialysis Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201603066DIPB
Record Dates: First submitted 2016-05-11; First posted 2016-05-25 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Patients on Dialysis
Keywords: Latent tuberculosis infection, dialysis
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dialysis group: Patient receiving long term dialysis
  Interventions: Other: Examination of latent TB by QuantiFERON-TB

INTERVENTIONS:
Other: Examination of latent TB by QuantiFERON-TB — Examination of latent TB by QuantiFERON-TB both QFT-plus QFT-GIT

SUMMARY:
In patients receiving long term dialysis, using new generation of QuantiFERON-TB Gold Plus can have less result variability in inter-experiment and serial follow up in comparing with QuantiFERON-TB Gold In-tube.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains one of the most important infectious diseases worldwide. According to the World Health Organization (WHO) estimates, there were 9 million new TB cases and 1.5 million related deaths in 2013. Future control strategies include early treatment for preventing transmission and treatment of latent TB infection (LTBI) for reducing reactivation. Patients with renal failure undergoing dialysis have increased risk of TB due to attenuated cellular immunity. For instance, their risk of developing active TB in the dialysis population is 7.8-25 times higher than that of the general population. However, TB diagnosis is usually delayed because of frequent extra-pulmonary manifestations. Thus, LTBI detection in this specific group is important.

Positive results of interferon-gamma release assays (IGRAs) and the exclusion of active TB are the current diagnostic bases of LTBI, which is a precursor of tuberculosis reactivation. However, recent reports show a high negative reversion rate of quantiFERON Gold In-tube (QFT-GIT), a kind of IGRA, in cohorts of health care workers (33% after 18 weeks) close TB contacts (35% after six months), and patients receiving long-term dialysis (46% after six months). This phenomenon questions the clinical significance of a single positive IGRA result. Increasing the IGRA threshold or doing serial follow-up to improve specificity have both been suggested but there is no comparison by the risk of TB development.

Therefore, increasing the accuracy and stability and then improving the rate of negative conversion from positive IGRA results are very important. Currently, new generation of QuantiFERON-TB Gold Plus includes two tubes for CD4 and CD8 T cells response, which can indicate TB immune response more specifically. The investigators applied this project to compare the performance of diagnosing LTBI by QuantiFERON-TB Gold Plus in comparing QuantiFERON-TB Gold In-tube.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20 years
* Receiving long term dialysis

Exclusion Criteria:

* Having tuberculosis previously

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis population
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
percentage of positive QFT | 1 week
  Compare the results of QFT-plus and QFT-GIT
percentage of positive QFT change | 1 week and 1 year
  Compare the change of the QFT-plus and QFT-GIT report by serial follow up

SECONDARY OUTCOMES:
percentage of occurrence of active TB | 2 year
  anticipated 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Select..., Taiwan

IPD SHARING:
Plan to Share IPD: Undecided